CLINICAL TRIAL: NCT00668759
Title: A Phase III Prospective, Randomized, Double-Blind, Active-Controlled, Multi-Center, Superiority Study of Vernakalant Injection Versus Amiodarone in Subjects With Recent Onset Atrial Fibrillation
Brief Title: A Phase III Superiority Study of Vernakalant vs Amiodarone in Subjects With Recent Onset Atrial Fibrillation
Acronym: AVRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Sheila Grant, VP Product Development and Product team leader, Vernakalant, Cardiome Pharma Corp.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VERI-305-AMIO
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial fib; AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vernakalant Injection:
  In one infusion line, subjects will receive a 10-minute infusion of vernakalant followed by a 15-minute observation period, followed by an additional 10-minute infusion of vernakalant if required (if the subject is still in AF). To maintain blinding, a 60-minute infusion of placebo (D5W) will be administered in a second infusion line, followed by a maintenance infusion of placebo for a minimum of an additional 60 minutes.
  Interventions: Drug: Vernakalant Injection
- 2 (Active Comparator): Amiodarone Injection:
  In one infusion line subjects will receive a 60-minute infusion of amiodarone followed by a maintenance infusion of amiodarone over an additional 60 minutes. To maintain blinding, a 10-minute infusion of placebo (normal saline) will be administered in a second infusion line, followed by a 15 minute observation period, followed by a 10 minute infusion of placebo if the subject is still in AF.
  Interventions: Drug: Amiodarone Injection:

INTERVENTIONS:
Drug: Vernakalant Injection — 10-minute infusion of 3 mg/kg vernakalant injection followed by a 15-minute observation period, followed by an additional 10-minute infusion of 2 mg/kg of vernakalant if required (if the subject is still in AF).
  Other Names: RSD1235; Kynapid
  Arms: 1
Drug: Amiodarone Injection: — 60-minute infusion of 5 mg/kg amiodarone followed by a maintenance infusion of 50 mg amiodarone over an additional 60 minutes (equivalent to approximately 15 mg/kg over 24 hrs).
  Other Names: Amiodarone; Cordarone
  Arms: 2

SUMMARY:
The primary objective of the study is to demonstrate the superiority of vernakalant injection over amiodarone injection in the conversion of atrial fibrillation (AF) to sinus rhythm (SR) within 90 minutes of the start of drug administration. The secondary objective is to compare the safety of vernakalant to amiodarone.

DETAILED DESCRIPTION:
This is a double-blind, active-controlled, double-dummy, multi-center, randomized trial in subjects with symptomatic AF of 3 to 48 hours duration.

Subjects will be randomized to receive vernakalant injection or amiodarone injection in a 1:1 ratio.

Safety will be assessed through the monitoring of adverse events, vital signs, continuous telemetry monitoring, 12-lead Holter monitoring, 12-lead ECGs, and laboratory tests.

At 2 hours after the start of infusion, electrical cardioversion may be performed or rate control medication may be administered. Class I and Class III antiarrhythmics are not to be administered for 24 hours after the start of infusion.

Subjects are to remain in the clinic for at least 6 hours after the start of infusion. Subjects will attend a follow-up visit at 7 (±2) days after treatment and will receive a follow-up telephone call at 30 (±3) days for assessment of serious adverse events, concomitant medications related to serious adverse events, and recurrence of AF.

All roles were blinded with the exception of each site's designated unblinded personnel who were responsible for randomization and preparation, dispensation and accountability of the study medication.

Expanded Access was not available through this protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Have symptomatic AF of 3 to 48 hours duration at baseline.
* Be eligible for cardioversion.
* Have adequate anticoagulation therapy for cardioversion in accordance with standard of practice as recommended by ACC/AHA/ESC guidelines [1].
* Be hemodynamically stable and have systolic blood pressure (BP) above 100 mmHg and less than 160 mmHg and diastolic BP less than 95 mmHg at screening and baseline.

Key Exclusion Criteria:

* Known or suspected prolonged QT or uncorrected QT interval of >440 msec as measured at screening on a 12 lead ECG, familial long QT syndrome, or previous torsades de pointes, ventricular fibrillation; or sustained ventricular tachycardia (VT).
* Symptomatic bradycardia, sick sinus syndrome, or ventricular rate less than 50 beats per minute (bpm) as documented by 12-lead ECG at screening.
* A QRS interval >140 msec.
* Atrial flutter.
* Significant valvular stenosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy or constrictive pericarditis.
* Documented previous episodes of second or third degree atrioventricular (AV) block.
* Had a myocardial infarction (MI), acute coronary syndrome or cardiac surgery within 30 days prior to entry into the study.
* Uncorrected electrolyte imbalance of serum potassium or magnesium. Both K+ and Mg2+ must be corrected prior to dosing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with conversion of atrial fibrillation to sinus rhythm within 90 minutes after the start of infusion. | Conversion of AF to SR for a minimum duration of one minute within 90 minutes after start of infusion.

SECONDARY OUTCOMES:
Time to conversion within 90 minutes after the start of infusion. | Time to conversion of AF to SR within 90 minutes after start of infusion.
Proportion of subjects with symptom relief at 90 minutes after the start of infusion. | Relief of AF symptoms 90 minutes after start of infusion.
EQ-5D quality of life assessment. | Assessment of quality of life 2 hours after start of infusion.
Monitoring of adverse events, vital signs, continuous telemetry monitoring, 12-lead Holter monitoring, 12-lead ECGs, and laboratory tests. | Specified safety assessments completed at specified time points throughout the study from Screening to Discharge, at the Day 7 visit, and at the Day 30 follow-up call.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Janota, MD, Principal Investigator — VFN III. interní klinika; Christian Torp-Pedersen, MD, Principal Investigator — Gentofte Amtssygehus - Kardiologisk afdeling; Rein Kolk, MD, Principal Investigator — Tartu University Hospital Heart Clinic; Etienne Aliot, MD, Principal Investigator — CHU de Nancy - Hopital Brabois, Service de Cardiologie; Stefan Hohnloser, MD, Principal Investigator — Johann Wolfgang Goethe Universitaet Med Klinik III - Kardiologie; Heikki Huikuri, MD, Principal Investigator — Oulu University Hospital - Dept of Internal Medicine; Piotr Ponikowski, MD, Principal Investigator — Osrodek Chorob Serca, Klinika Kardiologii, IV Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej we Wroclawiu; Steen Juul-Moller, MD, Principal Investigator — Universitetssjukhuset MAS
Locations (100):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital Cardiology Research, Hobart, Tasmania
  - Launceston General Hospital Cardiac Research Unit, Launceston, Tasmania
  - Royal Perth Hospital Emergency Research, Perth, Western Australia
- Canada (7):
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Centre Hopitalier de L'Universite de Montreal - Hotel Dieu, Montreal, Quebec
  - McGill University Health Center The Montreal General Hospital, Montreal, Quebec
  - Centre de santé et de services sociaux du Sud de Lanaudière - Hôpital Pierre-Le Gardeur, Terrebonne, Quebec
- Czechia (12):
  - Mestrska nemocnice Caslav, Čáslav
  - Nemocnice Kroměříž, Kroměříž
  - Nemocnice Kutna Hora s.r.o. Interni Oddeleni, Kutná Hora
  - Nemocnice Decin Internal Medicine, Nove Město
  - Fakultní nemocnice v Motole, KAR, Prague
  - Ustredni vojenska nemocnice Koronarni jednotka, Prague
  - VFN - III. Interni Klinika, Prague
  - Oblastni nemocnice Pribram Interni Oddeleni, Příbram
  - Nemocnice v Semilech Interní oddělení, Semily
  - Nemocnice Slaný Interní oddělení, Slaný
  - Nemocnice Tabor, Tábor
  - Uherskohradistska nemocnice, Uherské Hradiste
- Denmark (5):
  - Gentofte Amtssygehus Kardiologisk afdeling, Hellerup
  - Herlev Amtssygehus, Kardiologisk, Herlev
  - Sygehus Vendsyssel Hjorring, Hjørring
  - Roskilde Amts Sygehus Køge, Køge
  - Regionshospitalet Silkeborg, Silkeborg
- Estonia (4):
  - Viimsi Hospital, Heart Clinic, Haabneeme
  - Pärnu Hospital Department of Cardiology, Pärnu
  - East Tallinn Central Hospital-Clinic of Cardiology, Tallinn
  - Tartu University Hospital Heart Clinic, Tartu
- Oulu University Hospital - Dept of Internal Medicine, Oulu, Finland
- France (4):
  - Hopital Trousseau - Service de Cardiologie, Chambray-lès-Tours
  - CHU de Nancy - Hopital Brabois - Service de Cardiologie, Nancy
  - Hôpital Lariboisiere, Paris
  - CHU de Strasbourg - Hopital Hautepierre - Service de Cardiologie, Strasbourg
- Germany (17):
  - Charite Campus Mitte, Med. Klinik und Poliklinik mit Schwerpunkt Kardiologie und Angiologie, Berlin
  - Campus Virchow-Klinikum, Charite - Universitaetsmedizin Berlin, Berlin
  - Herzzentrum Brandenburg in Bernau Innere Medizin, Bernau
  - Universitätsklinikum Bonn, Med. Klinik und Poliklinik II, Bonn
  - Klinikum der Universität Köln, Medizinische Klinik III, Cologne
  - Johann Wolfgang Goethe Universitaet Med Klinik III - Kardiologie, Frankfurt
  - Universitatsklinikum Gottingen, Herzzentrum, Göttingen
  - Martin-Luther Universitat Halle, Med. Klinik und Poliklinik III- Fachrichtung Kardiologie, Halle
  - Klinik Hamburg Bambek Kardiologie, Hamburg
  - Medizinisches Versorgungszentrum Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Medizinische Klinik, Klinikum Hannover Nordstadt, Hanover
  - Ambulantes Herzzentrum Kassel Innere Medizin, Kassel
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Carl-von Basedow-Klinikum Merseburg, Merseburg
  - Klinikum Pirna GmbH, Innere Medizin II, Kardiologie, Pirna
  - Krankenhaus Reinbek, St. Adolf-Stift, Reinbek
  - Robert-Bosch-Krankenhaus, Abt. Kardiologie / Pulmologie, Stuttgart
- Latvian Center of Cardiology, P. Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (3):
  - Kaunas Medical University Hospital - Department of Cardiology, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic - Center of Cardiology and Angiology, Vilnius
- Netherlands (7):
  - WCN - Department of Cardiology Rijnstate Ziekenhuls, Arnhem
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Groene Hart Zeikenhhaus, Gouda
  - WCN - Bethesda ziekenhuis, Hoogeveen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - WCN - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - WCN - St. Franciscus Gasthuis, Rotterdam
- Poland (12):
  - Oddzial Kardiologiczny Wielospecjalityczny Szpital Miejski im., Bydgoszcz
  - Szpital Miejski im. J. Brudzinskiego Oddzial Kardiologii, Gdynia
  - Klinika Chorob Wewnetrznych z Oddzialem Farmakologii Klinicznej i Terapii Monitorowanej, Lodz
  - Oddział Internistyczno-Kardiologiczny Samodzielny Publiczny Szpital Wojewódzki im. Jana Bożego w Lublinie, Lublin
  - Okregowy Szpital Kolejowy w Lublinie Samodzielny, Lublin
  - Oddzial Kardiologii Inwazyjnej Szpital Specjalistyczny im. E.Szczeklika w Tarnowie, Tarnów
  - Oddział Kardiologiczno-Internistyczny Specjalistyczny Szpital Miejski im. Mikołaja Kopernika, Torun
  - Specjalistyczny Szpital Miejski im. Mikołaja Kopernika, Torun
  - III Klinika Chorob Wewnetrznych i Kardiologii, Warsaw
  - Wojskowy Instytut Medyczny, CSK MON, Warsaw
  - Klinika Kardiologii Zachowawczej Centralny Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji w Warszawie, Warsaw
  - Osrodek Chorob Serca, Klinika Kardiologii, 4 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny, Wroclaw
- Serbia (4):
  - Clinical Center of Serbia, Institute of CV Diseases, Belgrade
  - "Dedinje" Cardiovascular Institute, Belgrade
  - Institute of Treatment and Reahabilitation 'Niska Banja', Niška Banja
  - Clinical Center Zemun, Dept. of Cardiology, Zemun
- Slovakia (8):
  - Middle Slovak Institute of Cardiovascular Diseases (SUSCCH), Banska Bysterica
  - NsP Prievidza so sidlom v Bojniciah, Bojnice
  - Slovensky ustav srdcovych a cevnych chorob, Bratislava
  - ICU, Hospital Lipt. Mikulas, Liptovský Mikuláš
  - FN - I. interna klinika, Nitra
  - Liva - Central Military Hospital, Ružomberok
  - Interna klinika FN Trnava, Fakultna nemocnica Trnava, Trnava
  - Internal Dep. Hospital Žilina, Žilina
- Sweden (3):
  - Universitetssjukhuset MAS, Malmo
  - Universityetssjukhuset, Orebro, Örebro
  - Akademiska Sjukhuset, Uppsala, Uppsala
- Ukraine (8):
  - Donetsk Regional Clinical Hospital, Donetsk
  - City Clinical Hospital #8, Kharkiv
  - City Clinical Hospital #1 Intensive Care Unit, Kiev
  - Kiev City Clinical Hospital No 5, Coronary Care Unit, Kiev
  - N.D. Strazhesko Institute of Cardiology Intensive Care Unit, Kiev
  - Lugansk First Clinical Multiprofile Hospital #1, Cardiology, Luhansk
  - Lviv Reg St Clinical Treat-and-Diagn Cardio. Centre Dept of Myocardial Infarction, Lviv
  - City Clinical Hospital #9 Dept of Arrhythmia, Odesa

REFERENCES:
- [Derived] Camm AJ, Capucci A, Hohnloser SH, Torp-Pedersen C, Van Gelder IC, Mangal B, Beatch G; AVRO Investigators. A randomized active-controlled study comparing the efficacy and safety of vernakalant to amiodarone in recent-onset atrial fibrillation. J Am Coll Cardiol. 2011 Jan 18;57(3):313-21. doi: 10.1016/j.jacc.2010.07.046. PMID 21232669